CLINICAL TRIAL: NCT01856413
Title: An Open, Prospective, Single Arm Study Investigating Efficacy and Safety of Human Hepatitis B Immunoglobulin Zutectra in Liver Transplanted Patients - the ZEUS Study
Brief Title: A Clinical Trial of Zutectra in Patients Who Recently Received a Liver Transplant
Acronym: ZEUS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biotest (Industry)
Collaborators: AMS Advanced Medical Services GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BT 987; 2012-002516-51 (EudraCT Number)
Record Dates: First submitted 2013-05-15; First posted 2013-05-17 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Hepatitis B
Keywords: Prevention; Hepatitis B virus re-infection; HBV-DNA negative; Liver transplantation
MeSH Terms: conditions — Hepatitis B | interventions — BT088 immunoglobulin, human; hepatitis B hyperimmune globulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Zutectra (Experimental): Subcutaneous injections of Zutectra up to 1,000 IU (2 ml) per week.
  Interventions: Drug: Zutectra

INTERVENTIONS:
Drug: Zutectra — Subcutaneous injections of Zutectra up to 1,000 IU (2 ml) per week.
  Other Names: Human hepatitis B Immunoglobulin; HBIg

SUMMARY:
Patients who receive liver transplantation for hepatitis B virus (HBV) induced liver failure require longterm therapy to prevent HBV reinfection of the transplanted liver. The approved preventative treatment is a combination of antihepatitis B immunoglobulin (HBIg) and oral antiviral medication. In the first 6 months after liver transplantation, patients receive treatment with intravenous HBIg to maintain blood antihepatitis B (antiHBs)antibody concentrations above 100 IU/L, the level considered safe for preventing hepatitis B reinfection.

Zutectra is an HBIg preparation for subcutaneous injection that is approved in the EU for the 'prevention of HBV reinfection in HBV DNA negative patients ≥ 6 months after liver transplantation for hepatitis B induced liver failure'. The purpose of this study is to show that earlier subcutaneous HBIg treatment with Zutectra after liver transplantation can prevent hepatitis B reinfection.

Treatment with subcutaneous HBIg (Zutectra) at home is manageable for the majority of patients and is more convenient for patients compared to intravenous treatment that must take place in the hospital setting.

Fourty patients will take part in the study at approximately 19 centres in UK, France, Italy and Spain. Patients who are eligible for the study will receive treatment with Zutectra for 24 weeks.

During the study, the safety and effectiveness of Zutectra will be assessed by checking for symptoms of hepatitis B related infection, as well as monitoring blood levels of antiHBs antibodies and hepatitis B surface antigen (HBsAg).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained prior to orthotopic liver transplantation (OLT) - not more than 3 months before OLT
* Historical evidence within the last 4 weeks that HBV-DNA is undetectable at time point of signature of Informed Consent
* Male and female patients (age 18-75 years)
* Patients with the diagnosis of liver failure with hepatitis B infection
* Patients undergoing liver transplantation or re-transplantation
* HBsAg negative on day 7 or on day 14 after OLT
* HBV-DNA undetectable at OLT
* Serum HBs antibody concentration on day 7 or on day 14 after OLT ≥ 400 IU/l
* Stable patient in a condition which in the opinion of the investigator would permit safe participation in the study
* Willingness to fill out patient diary

Exclusion Criteria:

* Re-transplantation due to viral recurrence
* Positive HIV or HCV test at time of transplantation
* HBV-DNA positive at OLT
* Patients having received organs from HBsAg positive donors
* Pregnancy or unreliable contraceptive measures or lactation period (females only)
* Known intolerance to immunoglobulins or comparable substances (e.g. vaccination reaction)
* Known intolerance to proteins of human origin
* Participation in another interventional clinical trial within 90 days before entering the study or during the study and/or previous participation in this study (except screening failures)
* Suspicion of drug and/or alcohol abuse
* Inability or lacking motivation to participate in the study
* Employee or direct relative of an employee of the CRO, the study site, or Biotest

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Trough levels of serum anti-HBs antibody concentrations | 24 weeks

SECONDARY OUTCOMES:
Hepatitis B related re-infections | 24 weeks
  The number of all patients with hepatitis B related infections will be assessed by monitoring of clinical signs, liver function and measurement of HBsAg and HBV-DNA.

OTHER OUTCOMES:
Adverse Events | 24 weeks
  The number of adverse events will be documented including safety laboratory parameters reported as AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Samuel, Professeur, Principal Investigator — Hospital Paul Brousse, Centre Hepato-Biliaire
Locations (16):
- France (2):
  - Hopital de la Croix Rousse, Lyon
  - Hôpital Paul Brousse, Villejuif
- Italy (9):
  - Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari, Bari
  - S. Orsola Hospital, Bologna
  - Azienda ospedaliera "G. Brutzu" di Cagliari, Cagliari
  - Azienda Ospedaliera Ospedale Niguarda Ca Granda-Chirurgia, Milan
  - Liver and Multivisceral Transplant Center, University of Modena and Reggio Emilia, Modena
  - Azienda Ospedialera Universitaria di Padova, Padua
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - Fondazione Policlinico Tor-Vergata U.O.C., Roma
  - Molinette Hospital, Torino
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital 12 de Octubre, Madrid
- United Kingdom (2):
  - University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital, Birmingham
  - King's College Hospital, London